CLINICAL TRIAL: NCT00960908
Title: RESOLUTE-KOREA Registry - Registry to Evaluate the Efficacy of Zotarolimus-eluting Stent
Brief Title: Registry to Evaluate the Efficacy of Zotarolimus-Eluting Stent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Hyo-Soo Kim, MD, PhD, Seoul National University Hospital
Other Study IDs: RESOLUTE-KOREA
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Artery Disease
Keywords: Zotarolimus; Drug eluting stent; Endeavor Resolute
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Resolute: Prospective recruitment of Resolute arm will start in March 2009
  Interventions: Device: Endeavor Resolute stents
- Endeavor: The retrospective recruiting period of Endeavor arm comprises a fixed 2-year time between January 2006 and December 2008. The patients, who were treated with Endeavor in that period, will be enrolled if they agree to participate in this study.
  Interventions: Device: Endeavor Sprint stent

INTERVENTIONS:
Device: Endeavor Resolute stents — 2nd generation ZES
  Other Names: Endeavor Resolute
  Groups: Resolute
Device: Endeavor Sprint stent — 1st generation ZES
  Other Names: Endeavor Sprint
  Groups: Endeavor

SUMMARY:
The objective of this study is to evaluate the safety and long-term effectiveness of coronary stenting with the zotarolimus eluting stent (ZES) and to determine clinical device and procedural success during commercial use of ZES.

The investigators will compare 2nd generation ZE (Endeavor resolute, active prospective arm) with 1st generation ZES (Endeavor Sprint, retrospective arm).

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the informed consent form.
* Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form.

Exclusion Criteria:

* There are no exclusion criteria for this registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 4000 patients derived from a population of patients receiving percutaneous coronary intervention for ischemic heart disease will be enrolled in the present registry.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (composite of cardiac death, non-fatal MI, target lesion revascularization) | 12 months

SECONDARY OUTCOMES:
In-stent & In-segment Late Loss | 9 months
Stent Thrombosis | 1 year
Target Vessel Failure (composite of cardiac death, MI, and TVR) | 12 months
Any death, cardiac death, MI, TLR, TVR | 1 year
Composite rate of cardiac death and any MI | 1 year
Composite rate of all death and any MI | 1 year
Composite rate of all death, any MI (Q-wave and non Q-wave) and any repeat revascularization | 1 year
Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy | 1 year
Clinical device and procedural success | During the health care facility stay

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (19):
- South Korea (19):
  - Hallym University Sacred Heart Hospital, Anyang
  - Yongnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonbuk National Univesity Hospital, Iksan
  - Inje University Ilsan Paik Hospital, Ilsan
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Gachon Kil Medical Center, Inchon
  - Inha University Hospital, Inchon
  - Gyeongsang National University Hospital, Jinju
  - Pusan National University Hospital, Pusan
  - Bundang CHA Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Gangbuk Samsung Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Seoul Boramae Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - St. Vincent's Hospital, Suwon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si